CLINICAL TRIAL: NCT05646134
Title: Effects of Repetitive Transcranial Magnetic Stimulation (rTMS) on Upper Extremity Motor Function in Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Raimondas Savickas, Professor, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: rTMS_1
Record Dates: First submitted 2022-10-25; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Stroke, Ischemic
Keywords: Stroke; Stroke rehabilitation; Repetitive transcranial magnetic stimulation
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low Frequency Experimental Group (Experimental): Participants in this Arm will receive 10 sessions of Low Frequency (1 Hz) rTMS Participants in this Arm will receive 10 sessions of High Frequency (10 Hz) rTMS
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- High Frequency Experimental Group (Experimental): Participants in this Arm will receive 10 sessions of High Frequency (10 Hz) rTMS
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Sham Stimulation Control Group (Sham Comparator): Participants in this Arm will receive 10 sessions of Sham rTMS
  Interventions: Device: Sham Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Repetitive transcranial magnetic stimulation (rTMS) is a form of non-invasive brain stimulation therapy that modulates brain excitability.
  Arms: High Frequency Experimental Group; Low Frequency Experimental Group
Device: Sham Transcranial Magnetic Stimulation — During Sham Transcranial Magnetic Stimulation the coil will be facing the wall making the stimulation inactive
  Arms: Sham Stimulation Control Group

SUMMARY:
This clinical trial aims to evaluate the effects of repetitive transcranial magnetic stimulation (rTMS) on upper extremity motor function in stroke patients. The main questions it seeks to answer are:

1. Whether repetitive transcranial magnetic stimulation (rTMS) has a positive effect on upper extremity motor function in stroke patients.
2. Which stimulation protocol (low frequency - LF or high-frequency - HF) has better outcomes for improving upper extremity motor function in stroke patients? Participants will receive 10 procedures of repetitive transcranial magnetic stimulation (rTMS) over two weeks. They will be randomly assigned into low-frequency, high-frequency rTMS groups or sham stimulation groups. Upper extremity motor function will be evaluated twice: before stimulation and 3-4 weeks after stimulation.

Researchers will compare sham stimulation to see if it has the same or better outcomes for improving upper extremity motor function in stroke patients than real rTMS.

DETAILED DESCRIPTION:
The aim of this clinical trial is to evaluate the effects of repetitive transcranial magnetic stimulation (rTMS) on upper extremity motor function in stroke patients. The main questions it aims to answer are:

1. Whether repetitive transcranial magnetic stimulation (rTMS) has a positive effect on upper extremity motor function in stroke patients.
2. Which stimulation protocol (low frequency - LF or high-frequency - HF) has better outcomes for improving upper extremity motor function in stroke patients? Participants will receive 10 procedures of repetitive transcranial magnetic stimulation (rTMS) over two weeks. They will be randomly assigned into low-frequency, high-frequency rTMS groups or sham stimulation groups. Upper extremity motor function will be evaluated twice: before stimulation and 3-4 weeks after stimulation by conducting Fugl Meyer Assessment for Upper Extremity, Box and Blog test, nine-hole peg test, and by measuring hand grip strength.

Researchers will compare experimental groups with sham stimulation to see if it has the same or better outcomes for improving upper extremity motor function in stroke patients than real rTMS.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic stroke of the middle cerebral artery, confirmed by instrumental tests (CT, MRI).
2. Acute hemiplegia/hemiparesis, hand motor deficit, muscle strength ≤ 4 points (as assessed by the Lovett scale).
3. Time after the stroke before inclusion in the study is no more than 1 month.
4. No severe deficit in cognitive functions.

Exclusion Criteria:

1. Patients with implanted ferromagnetic or other metal devices sensitive to a magnetic field in the head or neck area; cochlear implants; implanted neurostimulators, pacemakers, or drug delivery pumps.
2. Complete aphasia or severe cognitive impairment.
3. Taking tricyclic antidepressants, neuroleptics, or benzodiazepines.
4. Previous skull fractures or other head injuries with loss of consciousness.
5. History of epilepsy or seizures.
6. Spasticity of the upper limb (Ashworth scale >2 b.).
7. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change of upper limb motor score in Fugl-Meyer Assessment | 7 weeks
  Fugl-Meyer test for Upper Extremity will be performed before and one month after 10 rTMS sessions. The minimum value of the Fugl-Meyer Assessment is 0 whereas the maximum value is 66 points. The higher the score the better the motor function of the upper extremity.
Change of Nine Hole Peg Test (9HPT) score | 7 weeks
  Nine Hole Peg Test (9HPT) will be performed before and one month after 10 rTMS sessions for measuring finger dexterity. During 9HPT a patient takes the pegs from a container, one by one, and places them into the holes on the board, as quickly as possible, using only the hand. The faster a patient finishes the test the better finger dexterity (measured by seconds).
Change of box and block test (BBT) score | 7 weeks
  Box and block test (BBT) will be performed before and one month after 10 rTMS sessions for measuring unilateral gross manual dexterity. During BBT a patient moves, one by one, the maximum number of blocks from one compartment of a box to another within 60 seconds. The more blocks are moved to another compartment the better the manual dexterity of the upper extremity.
Change of hand grip strength | 7 weeks
  Hand grip strength will be measured in kilograms using a dynamometer before and one month after 10 rTMS sessions. The higher the score the stronger the forearm muscles.

SECONDARY OUTCOMES:
Change of Functional Independence Measure (FIM) test score. | 7 weeks
  Functional Independence Measure (FIM) will be performed before and one month after 10 rTMS sessions. The minimum value of FIM is 18 whereas the maximum value is 126. The higher the score the better functional independence.

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania